CLINICAL TRIAL: NCT07065773
Title: An Open Label Study to Investigate the Safety and Tolerability of Trichostatin A in Patients With Mild to Severe Onychomycosis
Brief Title: Safety, Tolerability and Efficacy of Trichostatin A in Patients With Mild to Severe Onychomycosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VTR-297-2201
Record Dates: First submitted 2025-06-05; First posted 2025-07-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Onychomycosis of Toenail
Keywords: Onychomycosis; Onychomycosis of Toenail; Trichophyton rubrum; Trichophyton mentagrophytes
MeSH Terms: conditions — Onychomycosis | interventions — trichostatin A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trichostatin A (Experimental)
  Interventions: Drug: Trichostatin A

INTERVENTIONS:
Drug: Trichostatin A — Topical Study Drug

SUMMARY:
This is a multicenter, open label study designed to evaluate the safety, tolerability, and efficacy of topically administered VTR-297 solution. The efficacy objectives of the study will be assessed using fungal culture testing, Neutral Red Staining (NRS) microscopy examination, and KOH microscopy examination after 4 weeks of treatment with VTR-297.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide signed and dated written voluntary informed consent.
* Adults with diagnosis of mild-to-severe DLSO/DSO affecting at least one great toenail.
* Positive microscopic examination with KOH for dermatophyte hyphae.
* Positive dermatophyte culture or mixed dermatophyte/Candida culture.

Exclusion Criteria:

* Presence of other toenail infection.
* Any disease or condition that may interfere with the evaluation including other conditions that affect the toenails or significant active tinea pedis.
* History of other significant chronic fungal disease, psoriasis, lichen planus or use of drug medications for those indications 6 months prior to screening and during the study.
* Participation in a previous clinical trial 3 months prior to screening or participation in a research study concurrent with this study.
* Current or planned pregnancy during the trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 24 weeks
  Subjects will be asked about AEs weekly during the evaluation phase and at every follow-up visit; descriptions of AEs will include, at a minimum: date of onset, date ended, severity, seriousness, relationship to the study drug, and outcome.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Vanda Investigational Site, Fremont, California
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, New Brighton, Minnesota
  - Vanda Investigational Site, Pflugerville, Texas
  - Vanda Investigational Site, Forest, Virginia

IPD SHARING:
Plan to Share IPD: No